CLINICAL TRIAL: NCT01624792
Title: Eicosapentaenoic Acid and Protein Modulation to Induce Anabolism in Chronic Obstructive Pulmonary Disease (COPD): Aim 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, PhD, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2012-0171
Record Dates: First submitted 2012-06-05; First posted 2012-06-21 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease; Muscle Wasting
Keywords: Protein metabolism; casein protein; EPA; Fish oil
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Muscular Atrophy | interventions — Olive Oil; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy older adults (Experimental): Healthy controls will receive each intervention (olive oil or fish oil with 3.5 g EPA+DHA) one time and for only one day per intervention .
  Interventions: Dietary Supplement: Olive oil; Dietary Supplement: Fish oil
- COPD patients (Experimental): COPD patients will receive one out of three possible interventions (olive oil or fish oil with 3.5 g EPA+DHA or fish oil and placebo with 2 g EPA+DHA) for 4 (+/- 7 days) weeks.
  Interventions: Dietary Supplement: Olive oil; Dietary Supplement: Fish oil; Dietary Supplement: Fish oil and placebo

INTERVENTIONS:
Dietary Supplement: Olive oil — Dose: 7.0 g/day (= 7 capsules/day).
Dietary Supplement: Fish oil — Dose: 7.0 g/day (= 7 capsules/day = 3.5g EPA+DHA/day).
Dietary Supplement: Fish oil and placebo — Dose: 7.0 g/day (= 4 capsules/day fish oil = 2.0g EPA+DHA/day and 3 capsules/day olive oil).
  Arms: COPD patients

SUMMARY:
Loss of muscle protein is generally a central component of weight loss in Chronic Obstructive Pulmonary Disease (COPD) patients. Gains in muscle mass are difficult to achieve in COPD unless specific metabolic abnormalities are targeted. The investigators recently observed that alterations in protein metabolism are present in normal weight COPD patients. Elevated levels of protein synthesis and breakdown rates were found in this COPD group indicating that alterations are already present before muscle wasting occurs. The investigators recently observed that in order to enhance protein anabolism, manipulation of the composition of proteins and amino acids in nutrition is required in normal-weight COPD. Intake of casein protein resulted into significant protein anabolism in these patients. The anabolic response to casein protein was even higher than after whey protein intake.

A substantial number of COPD patients, underweight as well as normal weight to obese, is characterized by an increased inflammatory response. This group failed to respond to nutritional therapy. Previous experimental research and clinical studies in cachectic conditions (mostly malignancy) indicate that polyunsaturated fatty acids (PUFA) are able to attenuate protein degradation by improving the anabolic response to feeding and by decreasing the acute phase response. Eicosapentaenoic acid (EPA) (in combination with docosahexaenoic acid (DHA)) has been shown to effectively inhibit weight loss in several disease states, however weight and muscle mass gain was not present or minimal.

Until now, limited research has been done examining muscle protein metabolism and the response to EPA and DHA supplementation in patients with COPD.

It is the investigator's hypothesis that supplementation of 2g/day EPA+DHA in COPD patients during 4 consecutive weeks will increase the muscle anabolic response to a high quality protein supplement as compared to a placebo, and supplementation of 3.5g/day EPA+DHA will increase the anabolic response even further. In the present study both the acute and chronic effects of EPA+DHA versus a placebo on muscle and whole body protein metabolism will be examined. The principal endpoint will be the extent of stimulation of net fractional muscle protein synthesis as this is the principal mechanism by which the effect of EPA+DHA on muscle anabolism can be measured. The endpoint will be assessed by isotope methodology which is thought to be the reference method.

DETAILED DESCRIPTION:
Specific aim 1: To test the hypothesis that supplementation of 3.5g EPA+DHA will increase the acute net fractional muscle protein synthesis more in COPD patients as compared to healthy controls in response to a high quality protein supplement.

Specific aim 2: To test the hypothesis that 3.5g/day EPA+DHA for 4 consecutive weeks induces a higher increase in net fractional muscle protein synthesis in response to a high quality protein supplement as compared to 2g/day EPA+DHA in COPD patients.

Therefore, to answer the specific aims in this study only the COPD subjects will undergo a 4-week intervention period.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria COPD subjects:

* Ability to walk, sit down and stand up independently
* Age 45 years or older
* Ability to lay in supine or elevated position for 8 hours
* Diagnosis of moderate to severe chronic airflow limitation, defined as measured forced expiratory volume in one second (FEV1) ≤ 70% of referen¬ce FEV1
* Clinically stable condition and not suffering from respiratory tract infection or exacerbation of their disease (defined as a combination of increased cough, sputum purulence, shortness of breath, systemic symptoms such as fever, and a decrease in FEV1 > 10% compared with values when clinically stable in the preceding year) at least 4 weeks prior to the study
* Shortness of breath on exertion
* Willingness and ability to comply with the protocol, including:

  * Refraining from alcohol consumption (24 h) and intense physical activities (72h) prior to each study visit
  * Adhering to fasting state from 10 pm ± 2h onwards the day prior to each study visit

Inclusion criteria healthy control subjects:

* Healthy male or female according to the investigator's or appointed staff's judgment
* Ability to walk, sit down and stand up independently
* Age 45 years or older
* Ability to lay in supine or elevated position for 8 hours
* No diagnosis of COPD and forced expiratory volume in one second (FEV1) > 80% of referen¬ce FEV1
* Willingness and ability to comply with the protocol, including:

  * Refraining from alcohol consumption (24 h) and intense physical activities (72h) prior to each study visit
  * Adhering to fasting state from 10 pm ± 2h onwards the day prior to each study visit

Exclusion Criteria:

* Any condition that may interfere with the definition 'healthy subject' according to the investigator's judgment (for healthy control group only)
* Established diagnosis of malignancy
* Established diagnosis of Diabetes Mellitus
* History of untreated metabolic diseases including hepatic or renal disorder
* Presence of acute illness or metabolically unstable chronic illness
* Recent myocardial infarction (less than 1 year)
* Any other condition according to the PI or study physicians would interfere with proper conduct of the study / safety of the patient
* BMI ≥ 40 kg/m2
* Dietary or lifestyle characteristics:

  * Use of supplements containing EPA+DHA 3 months prior to the first test day Use of protein or amino acid containing nutritional supplements within 5 days of first study day
  * Current alcohol or drug abuse
* Indications related to interaction with study products:

  * Known allergy to milk or milk products
  * Known hypersensitivity to fish and/or shellfish, Swanson EFAs Super EPA Fish oil or any of its ingredients, Swanson EFAs Certified Organic Extra Virgin Olive oil or any of its ingredients
* Contraindications to biopsy procedure:

  * Platelet count (PLT) < 100,000
  * History of hypo- or hyper-coagulation disorders including use of a Coumadin derivative, history of deep venous thrombosis (DVT), or pulmonary embolism (PE) at any point in lifetime
  * Currently taking anti-thrombotics and cannot stop for 7 days (i.e. medical indication)
  * Allergy to local anesthetic
* Use of long-term oral corticosteroids or short course of oral corticosteroids in the preceding month before enrollment
* Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-10-25 (Actual); Primary Completion 2016-06-29 (Actual); Study Completion 2016-06-29 (Actual)

PRIMARY OUTCOMES:
Fractional muscle protein synthesis and breakdown rate (FSR and FBR) of mixed muscle protein (%/h) and net fractional muscle protein synthesis (nFSR = FSR - FBR) | Acutely before and after 4 hours of feeding and the change after 4 weeks of EPA+DHA or placebo supplementation
  On the study days the primary outcome measure is determined acutely before and after 4 hours of feeding and after intake of either the 3.5 g EPA+DHA, a placebo or 2.0 g EPA+DHA (last category only applicable to COPD group). After study day 1 COPD patients undergo a 4-week intervention period of daily EPA+DHA or placebo supplementation and on their return visit (2nd study day) the primary outcome measure is determined again.

SECONDARY OUTCOMES:
Net whole body protein synthesis (whole body protein synthesis and breakdown rate) | Acutely before and after 4 hours of feeding and the change after 4 weeks of EPA+DHA or placebo supplementation
  On the study days the primary outcome measure is determined acutely before and after 4 hours of feeding and after intake of either the 3.5 g EPA+DHA, a placebo or 2.0 g EPA+DHA (last category only applicable to COPD group). After study day 1 COPD patients undergo a 4-week intervention period of daily EPA+DHA or placebo supplementation and on their return visit (2nd study day) the primary outcome measure is determined again.
Whole body myofibrillar protein breakdown rate | Acutely before and after 4 hours of feeding and the change after 4 weeks of EPA+DHA or placebo supplementation
  On the study days the primary outcome measure is determined acutely before and after 4 hours of feeding and after intake of either the 3.5 g EPA+DHA, a placebo or 2.0 g EPA+DHA (last category only applicable to COPD group). After study day 1 COPD patients undergo a 4-week intervention period of daily EPA+DHA or placebo supplementation and on their return visit (2nd study day) the primary outcome measure is determined again.
Glutathione turnover | Acutely before and after 4 hours of feeding and the change after 4 weeks of EPA+DHA or placebo supplementation
  On the study days the primary outcome measure is determined acutely before and after 4 hours of feeding and after intake of either the 3.5 g EPA+DHA, a placebo or 2.0 g EPA+DHA (last category only applicable to COPD group). After study day 1 COPD patients undergo a 4-week intervention period of daily EPA+DHA or placebo supplementation and on their return visit (2nd study day) the primary outcome measure is determined again.
Body composition | On study day 1 and the change from study day 1 on study day 2
  Body composition as measured by Dual-Energy X-ray Absorptiometry. Determined on study day 1 and after 4 weeks on study day 2 for COPD patients.
Skeletal and respiratory muscle strength and fatigue | On study day 1 and the change from study day 1 on study day 2
  Determined on study day 1 and after 4 weeks on study day 2 for COPD patients.
Inflammatory profile (CRP, IL6, IL1b, TNFα, IL8 and IL10) | On study day 1 and the change from study day 1 on study day 2
  Determined on study day 1 and after 4 weeks on study day 2 for COPD patients.
Other plasma products | On study day 1 and the change from study day 1 on study day 2
  Insulin, glucose, urea, cortisol, lactate, blood fatty acid profile (EPA, DHA, arachidonic acid, protectins and resolvins). Some of the parameters are measured on a single occasion and others are measured repeatedly during 10 hours on each study day (e.g. insulin and glucose). Determined on study day 1 and after 4 weeks on study day 2 for COPD patients.
Oxidative capacity | On study day 1 and 2
  Oxidative capacity, including peroxisome proliferator-activated receptor (PPAR) and muscle fiber typing. Determined before and after 4 hours of feeding.
Molecular markers (mTOR) of muscle wasting | On study day 1 and the change from study day 1 on study day 2

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Engelen, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University, College Station, Texas, United States

REFERENCES:
- [Derived] Engelen MPKJ, Kirschner SK, Coyle KS, Argyelan D, Neal G, Dasarathy S, Deutz NEP. Sex related differences in muscle health and metabolism in chronic obstructive pulmonary disease. Clin Nutr. 2023 Sep;42(9):1737-1746. doi: 10.1016/j.clnu.2023.06.031. Epub 2023 Jul 26. PMID 37542951
- [Derived] Engelen MPKJ, Jonker R, Sulaiman H, Fisk HL, Calder PC, Deutz NEP. omega-3 polyunsaturated fatty acid supplementation improves postabsorptive and prandial protein metabolism in patients with chronic obstructive pulmonary disease: a randomized clinical trial. Am J Clin Nutr. 2022 Sep 2;116(3):686-698. doi: 10.1093/ajcn/nqac138. PMID 35849009